CLINICAL TRIAL: NCT04083274
Title: Efficacy of Ultrasound-Guided Erector Spinae Plane Block for Pain Management Following Upper Extremity Surgery
Brief Title: Ultrasound-Guided Erector Spinae Plane Block Following Upper Extremity Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Primary researcher, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Medipol Hospital 4
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Upper Extremity Problem
Keywords: Upper extremity surgery; Postoperative pain management; Erector spina plane block

STUDY DESIGN:
Intervention Model Description: There are two models for this study. The first group is erector spinae plane block group. The second one is sham block group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patient, the investigator and the anesthesiologist who performs postoperative pain evaluation will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group E = ESPB group (Active Comparator): In group E, ESPB will be performed. US probe will be placed longitudinally 2-3 cm lateral to the T2 transvers process. Erector spinae muscle will be visualized on the hyperechoic transverse process. The block needle will be inserted caudo-cranial direction and then for correction of the needle 5 ml saline will be enjected deep into the erector spina muscle fascia. Following confirmation of the correct position of the needle 30 ml %0.25 bupivacaine will be administered for block.
  Interventions: Other: Erector spinae plane block (Group E)
- Group S = Sham block group (Sham Comparator): In group S, sham block will be performed. US probe will be placed longitudinally 2-3 cm lateral to the T2 transvers process. Erector spinae muscle will be visualized on the hyperechoic transverse process. The block needle will be inserted caudo-cranial direction and then for correction of the needle 5 ml saline will be enjected deep into the erector spina muscle fascia. Following confirmation of the correct position of the needle 30 ml normal saline will be administered for block.
  Interventions: Other: Sham block group (Group S)

INTERVENTIONS:
Other: Erector spinae plane block (Group E) — Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. Postoperative patient evaluation will be performed by an anesthesiologist blinded to the procedure.
  Postoperative pain assessment will be performed using the VAS score (0 = no pain, 10 = the most severe pain felt). The VAS scores at rest and during cough will be recorded at postoperative 1, 2, 4, 8, 16, 24 and 48 hours. If the VAS score will be ≥ 4, 0.5 mg/ kg meperidine IV will be administered. Sedation level will be assessed with a 4-point sedation scale (0 = awake, eyes open, 1 = sleepy but responding to verbal stimulus, 2 = sleepy and hard to evoke, 3 = sleepy, not aroused by shaking). The first time of the use of rescue analgesic, intraoperative and postoperative opioid consumption, side effects such as nausea, vomiting, itching and block related complications will be recorded.
  Arms: Group E = ESPB group
Other: Sham block group (Group S) — Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. Postoperative patient evaluation will be performed by an anesthesiologist blinded to the procedure.
  Postoperative pain assessment will be performed using the VAS score (0 = no pain, 10 = the most severe pain felt). The VAS scores at rest and during cough will be recorded at postoperative 1, 2, 4, 8, 16, 24 and 48 hours. If the VAS score will be ≥ 4, 0.5 mg/ kg meperidine IV will be administered. Sedation level will be assessed with a 4-point sedation scale (0 = awake, eyes open, 1 = sleepy but responding to verbal stimulus, 2 = sleepy and hard to evoke, 3 = sleepy, not aroused by shaking). The first time of the use of rescue analgesic, intraoperative and postoperative opioid consumption, side effects such as nausea, vomiting, itching and block related complications will be recorded
  Arms: Group S = Sham block group

SUMMARY:
Postoperative pain is important following upper extremity surgery. Postoperative effective pain treatment provides early mobilization and shorter hospital stay.Ultrasound (US)-guided brachial plexus blocks such as interscalen, axillary, infraclavicular and supraclavicular block are usually performed.

The US-guided erector spina plane block (ESPB) is a novel interfacial plan block defined by Forero et al. Local anesthetic injection is administrated into the deep fascia of erector spinae. ESPB provides thoracic analgesia at T5 level, abdominal analgesia at T7-9 level, and lumbar analgesia at T10-12, L3 levels. There are a few case reports about the efficacy of ESPB for acute and chronic shoulder pain. However, there are no randomized clinical studies. The aim of this study is to evaluate the efficacy of the US-guided ESPB for postoperative analgesia management after upper extremity surgery.

DETAILED DESCRIPTION:
Postoperative pain is an important issue in patients underwent upper extremity surgery. Pain causes a few problems; discomfortable patients, negative outcomes and longer rehabilitation. Postoperative effective pain treatment provides early mobilization and shorter hospital stay, thus complications due to hospitalization such as infection and thromboembolism may be reduced. Various techniques may be used for postoperative pain treatment. Opioids are one of the most preferred drugs among the analgesic agents. Parenteral opioids are generally performed for patients after surgery. However opioids have undesirable adverse events such as nausea, vomiting, itching, sedation and respiratory depression (opioid-related adverse events).

Various methods may be performed to reduce the use of systemic opioids and for effective pain treatment following arthroscopic shoulder surgery. Ultrasound (US)-guided brachial plexus blocks such as interscalen, axillary, infraclavicular and supraclavicular block are commonly used.

US-guided interfascial plane blocks have been used increasily due to the advantages of ultrasound in anesthesia practice. The US-guided erector spina plane block (ESPB) is a novel interfacial plan block defined by Forero et al. at 2016. The ESPB contains a local anesthetic injection into the deep fascia of erector spinae. This area is away from the pleural and neurological structures and thus minimizes the risk of complications due to injury. Visualization of sonoanatomy with US is easy, and the spread of local anesthesic agents can be easily seen under the erector spinae muscle. Thus, analgesia occurs in several dermatomes with cephalad-caudad way. Cadaveric studies have shown that the injection spreads to the ventral and dorsal roots of the spinal nerves. ESPB provides thoracic analgesia at T5 level, abdominal analgesia at T7-9 level, and lumbar analgesia at T10-12, L3 levels. To the best of our knowledge, there have been a few case reports about the efficacy of ESPB for acute and chronic shoulder pain. There are no randomized clinical studies, yet.

The aim of this study is to evaluate the efficacy of the US-guided ESPB for postoperative analgesia management after underwent upper extremity surgery. The primary aim is to compare perioperative and postoperative opioid consumption and the secondary aim is to evaluate postoperative pain scores (VAS), adverse effects related with opioids (allergic reaction, nausea, vomiting).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for upper extremity surgery under general anesthesia

Exclusion Criteria:

* history of bleeding diathesis,
* receiving anticoagulant treatment,
* known local anesthetics and opioid allergy,
* infection of the skin at the site of the needle puncture,
* pregnancy or lactation,
* patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | Change from baseline opioid consumption at postoperative 1, 2, 4, 8, 16, 24 and 48 hours
  The primary aim is to compare perioperative and postoperative opioid consumption

SECONDARY OUTCOMES:
Pain scores (Visual analogue scores-VAS) | Changes from baseline pain scores at postoperative 1, 2, 4, 8, 16, 24 and 48 hours.
  Postoperative pain assessment will be performed using the VAS score (0 = no pain, 10 = the most severe pain felt). The VAS scores at rest and during cough will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not plan to share IPD

REFERENCES:
- [Background] Forero M, Rajarathinam M, Adhikary SD, Chin KJ. Erector spinae plane block for the management of chronic shoulder pain: a case report. Can J Anaesth. 2018 Mar;65(3):288-293. doi: 10.1007/s12630-017-1010-1. Epub 2017 Nov 13. PMID 29134518
- [Background] Selvi O, Tulgar S, Ozer Z. Case Report Presentation of Ultrasound-guided Erector Spinae Plane Block in Shoulder Surgery: Three Patients and Two Different Results. Cureus. 2018 Nov 3;10(11):e3538. doi: 10.7759/cureus.3538. PMID 30648071
- [Background] Wiegel M, Moriggl B, Schwarzkopf P, Petroff D, Reske AW. Anterior Suprascapular Nerve Block Versus Interscalene Brachial Plexus Block for Shoulder Surgery in the Outpatient Setting: A Randomized Controlled Patient- and Assessor-Blinded Trial. Reg Anesth Pain Med. 2017 May/Jun;42(3):310-318. doi: 10.1097/AAP.0000000000000573. PMID 28257388